CLINICAL TRIAL: NCT03079115
Title: Efficacy of Two Different Doses of Atorvastatin for Prevention of Periprocedural Ischemic Brain Damage in Chinese Patients Undergoing Carotid Artery Stenting (CAS)
Brief Title: High Dose Atorvastatin for Preventing Periprocedural Ischemic Brain Damage During Carotid Artery Stenting
Acronym: PICAS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Hospital (Other Government)
Responsible Party: Principal Investigator, Jun Lu, Attending Physician; MD, Beijing Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 121-2016006
Record Dates: First submitted 2017-03-06; First posted 2017-03-14 (Actual); Last update posted 2020-04-09 (Actual); Status verified 2020-04

CONDITIONS: Carotid Artery Stenosis
Keywords: Atorvastatin
MeSH Terms: conditions — Carotid Stenosis | interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-dose Atorvastatin Arm (Active Comparator): High dose Atorvastatin (80 mg QD from 3 days before to 3 days after carotid artery stenting, thereafter conventional dose of Atorvastatin with 20mg QD until 30 days after CAS)
  Interventions: Drug: High-dose Atorvastatin
- Conventional-dose Atorvastatin Arm (Other): Conventional dose Atorvastatin (20mg QD from 3 days before to 30 days after CAS)
  Interventions: Drug: Conventional-dose Atorvastatin

INTERVENTIONS:
Drug: High-dose Atorvastatin — high-dose Atorvastatin (80 mg QD from 3 days before to 3 days after CAS, and thereafter 20mg QD until 30 days after CAS)
  Other Names: Lipitor
  Arms: High-dose Atorvastatin Arm
Drug: Conventional-dose Atorvastatin — conventional-dose Atorvastatin(20 mg QD from 3 days before to 30 days after CAS).
  Other Names: Lipitor
  Arms: Conventional-dose Atorvastatin Arm

SUMMARY:
The purpose is to test whether a short-term, high-dose atorvastatin treatment (80mg once a daily (QD) from 3 days before to 3 days after CAS, then 20 mg QD until 30 days after CAS) is superior to conventional-dose atorvastatin treatment (20 mg QD from 3 days before to 30 days after CAS), in terms of efficacy for prevention of periprocedural ischemic brain damage in Chinese patients undergoing CAS.

DETAILED DESCRIPTION:
Chinese patients with carotid stenosis scheduled for selective CAS will be randomized into two groups. The High-dose Atorvastatin group will receive Atorvastatin 80 mg QD from 3 days before to 3 days after CAS, then 20 mg QD until 30 days after CAS, while the Conventional-dose Atorvastatin group will receive Atorvastatin 20 mg QD from 3 days before to 30 days after CAS. All patients will receive cerebral diffusion-weighted (DW)-MRI within 7 days before CAS. Then, they will also receive repeated DW-MRI within 5 days after CAS. Efficacy for prevention of periprocedural ischemic brain damage of the two different Atorvastatin treatments will be compared, in terms of periprocedural incidence of transient ischemic attack (TIA)/ ischaemic stroke or new ischemic lesions on cerebral DW-MRI.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 50% stenosis of internal carotid artery in symptomatic patients; or ≥ 70% stenosis of internal carotid artery in asymptomatic patients
* received statin therapy for ≥ 2weeks before inclusion

Exclusion Criteria:

* nonatherosclerotic carotid disease (dissection, radiation-induced stenosis)
* received endovascular procedure within 30 days before inclusion
* CAS during the procedure of urgent endovascular therapy for acute ischaemic stroke
* need for oral anticoagulant therapy
* high risk of bleeding or contraindications to antiplatelet therapy (eg: platelet count <70 X 109/L)
* active hepatic disease or hepatic dysfunction, or aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 1.5 upper normal limit
* myopathy or increased creatine kinase (CK) > 2 upper normal limit
* renal failure with serum creatinine (Scr) > 3 mg/dl or 264μmol/L
* unable to undergo MRI because of claustrophobia or pacemaker
* pregnancy, lactation, or child bearing potential women without any effective contraception

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2017-08-21 (Actual); Primary Completion 2020-04-30 (Estimated); Study Completion 2020-04-30 (Estimated)

PRIMARY OUTCOMES:
brain damage | 30 days
  composite incidence of new ischemic lesion on post-CAS cerebral DW-MRI, TIA or ischaemic stroke within 30 days after CAS

SECONDARY OUTCOMES:
ischemic brain damage-1 | within 5 days
  incidence of new ischemic lesion on post-CAS DW-MRI
ischemic brain damage-2 | within 5 days
  number of new lesions on post-CAS DW-MRI
ischemic brain damage-3 | within 5 days
  incidence of new lesion > 5 mm on post-CAS DW-MRI
ischemic brain damage-4 | 30 days
  composite incidence of TIA or ischaemic stroke within 30 days after CAS
death, any stroke, or myocardial infarction | 30 days
  composite incidence of death, any stroke, or myocardial infarction within 30 days after CAS

CONTACTS AND LOCATIONS:
Overall Officials: Jun Lu, M.D., Principal Investigator — Beijing Hospital
Locations (1):
- Beijing Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang H, Wang J, Qi P, Yang X, Chen K, Hu S, Liu E, Zhang S, Gao Q, Li R, Lu J, Deng G, Wang D. A single-center pilot randomized controlled trial of atorvastatin loading for preventing ischemic brain damage after carotid artery stenting. Front Aging Neurosci. 2022 Dec 23;14:1066316. doi: 10.3389/fnagi.2022.1066316. eCollection 2022. PMID 36620770
- [Derived] Wang H, Wang J, Lu J, Wang D. Effects of High Dose of Atorvastatin for Preventing Periprocedural Ischemic Brain Damage in Patients Undergoing Carotid Artery Stenting (PICAS) in China: A Randomized Controlled Clinical Trial. Front Neurol. 2020 Aug 25;11:937. doi: 10.3389/fneur.2020.00937. eCollection 2020. PMID 32982944